CLINICAL TRIAL: NCT04913870
Title: Impact of Angiotensin Receptor Blockers in Aortic Stenosis - a Randomized Controlled Trial
Brief Title: Angiotensin Receptor Blockers in Aortic Stenosis
Acronym: ARBAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marie-Annick Clavel, Full Professor, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21617
Record Dates: First submitted 2021-05-03; First posted 2021-06-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-03

CONDITIONS: Aortic Stenosis; Aortic Valve Stenosis
Keywords: Angiotensin II Receptor Blockers; Left ventricular remodeling; Valvular heart disease; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Remodeling; Heart Valve Diseases | interventions — Angiotensin Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiotensin Receptor Blockers (Experimental): Angiotensin Receptor Blockers will be given orally once a day for 2 years.
  Interventions: Drug: Angiotensin Receptor Blockers
- Placebo (Placebo Comparator): Participants will receive a matched placebo orally once a day for 2 years.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Angiotensin Receptor Blockers — Angiotensin Receptor Blockers treatment for 2 years.
  Arms: Angiotensin Receptor Blockers
Other: Placebo — Placebo administration for 2 years.
  Arms: Placebo

SUMMARY:
This study is intended to investigate the effect of angiotensin receptor blockers (ARBs) on mild-to-moderate aortic stenosis.

DETAILED DESCRIPTION:
Studies support the concept that activation of the renin-angiotensin system may be involved in the progression of valve stenosis and myocardial fibrosis in aortic stenosis. Furthermore recent studies have shown that renin-angiotensin system medication may slow down aortic stenosis progression rate and left ventricle remodeling.

Thus the present study is a randomized control trial to test the efficacy of the angiotensin receptor blocker (ARB) to slow down aortic stenosis progression and left ventricular remodeling/dysfunction in patients with mild-to-moderate aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate aortic stenosis (peak aortic jet velocity ≥2.5 and <4m/s)
* Normal left ventricular ejection fraction (i.e. ≥50%)
* Systolic blood pressure >110 mmHg
* Diastolic blood pressure >70 mmHg

Exclusion Criteria:

* More than mild aortic or mitral regurgitation, or mitral stenosis
* Current use or documented indication for renin-angiotensin system medication or Aliskiren
* Known allergy or intolerance to angiotensin II receptor blockers (ARBs)
* Alzheimer, dementia or known non-compliant patient
* Renal dysfunction (glomerular filtration rate <30ml/min/1.73m2)
* Chronic hyperkalemia
* Diagnosed hepatic failure, cirrhosis, hepatitis or history of hepatic impairment
* Newly diagnosed (<2 months) or poorly controlled diabetes
* Pre-existing obstructive coronary artery disease with CCS III-IV angina or recent myocardial infarction (<3 months)
* Pregnant or lactating women
* Patients unable to read, understand or sign research consent

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in the anatomic progression of aortic stenosis | Baseline, 2 years
  Aortic valve calcification (measured by MDCT)

SECONDARY OUTCOMES:
Change in peak aortic jet velocity | Baseline, 2 years
  peak aortic jet velocity (Echocardiography)
Change in aortic valve area | Baseline, 2 years
  Aortic valve area (Echocardiography)
Change in left ventricular (LV) dimension | Baseline, 2 years
  LV dimension (Echocardiography, MRI)
Change in left ventricular (LV) mass | Baseline, 2 years
  LV mass (Echocardiography, MRI)
Change in left ventricular (LV) fibrosis | Baseline, 2 years
  LV Fibrosis (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Annick Clavel, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (2):
- CRIUCPQ, Québec, Quebec, Canada
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No